CLINICAL TRIAL: NCT02561494
Title: Postoperative Analgesic Effect of Nefopam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Doctor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nefo_stomach op
Record Dates: First submitted 2015-08-02; First posted 2015-09-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nefopam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Control (Placebo Comparator): Intravenous normal saline 2 ml is given slowly as a placebo before the anesthesia induction and after finishing anesthesia.
  Interventions: Drug: Saline
- Nefopam (Experimental): Intravenous nefopam 20 mg is given slowly before the anesthesia induction and after finishing anesthesia.
  Interventions: Drug: Nefopam

INTERVENTIONS:
Drug: Nefopam
  Arms: Nefopam
Drug: Saline
  Arms: Control

SUMMARY:
Nefopam will be administered to the patients undergoing laparoscopic gastrectomy under the total intravenous anesthesia (TIVA).

The investigators will evaluate whether the nefopam can decrease the total amount of remifentanil administered during the operation, which will reduce the acute opioid tolerance and following consumption of fentanyl during postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Early or advanced gastric cancer

Exclusion Criteria:

* Refusal
* Use of preoperative analgesic drugs
* Pregnancy
* Recurred gastric cancer
* Seizure
* Cardiac disease
* Monoamine oxidase inhibitor
* Urologic disease
* Previous intrabdominal surgery
* Body mass index > 30 or < 16

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change of the administered fentanyl dose from postoperative 6 h to postoperative 5 day | postoperative 6 h, postoperative 1 day, postoperative 2 day, postoperative 3 day, postoperative 5 day

SECONDARY OUTCOMES:
Change of the pain score from postoperative 6 h to postoperative 5 day | postoperative 6 h, postoperative 1 day, postoperative 2 day, postoperative 3 day, postoperative 5 day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea